CLINICAL TRIAL: NCT03764137
Title: Imaging with [89Zr]Panitumumab-PET/MRI in Patients with Newly Diagnosed Colorectal Cancer
Acronym: Panitumumab
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was not able to enroll any subjects
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Suzanne E. Lapi, PhD, Director Cyclotron Facility, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 300002089
Record Dates: First submitted 2018-11-01; First posted 2018-12-04 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [89Zr]Panitumumab-PET/MRI patients (Experimental): All study patients will receive [89Zr]Panitumumab-PET/MRI imaging.
  Interventions: Drug: [89Zr]Panitumumab PET-MRI

INTERVENTIONS:
Drug: [89Zr]Panitumumab PET-MRI — All patients entered into the study will have [89Zr]Panitumumab-PET/MRI imaging.

SUMMARY:
This clinical study will investigate the utility of PET imaging with [89Zr]Panitumumab for imaging of EGFR expression in newly diagnosed colon cancer patients to assess lymph node involvement. If promising, this data will be used to design larger trials.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 19 years of age.
* Diagnosis of colon cancer
* Scheduled to undergo surgical resection

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Inability to lie still for the imaging study
* Weight over 350 lbs., due to the scanner bore size
* Contraindication for MRI study (e.g. non-removable metal implants or certain tattoos)
* Inability to receive Omnipaque (iohexol) iodinated contrast
* Inability to receive glucagon
* Inability to receive Eovist (gadoxetate disodium) gadolinium based contrast agent
* Allergy to contrast imaging agents
* Finding or suspicion of distant metastases on CT

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Image Quality | 12 months
  Diagnostic image quality of [89Zr]Panitumumab PET imaging in patients with newly diagnosed colon cancer with nodal involvement. Standardized Uptake Values (SUVs) will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Lapi, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No